CLINICAL TRIAL: NCT04201665
Title: Uterine Electromyography for Estimation of Uterotonic Efficiency for Postpartum Hemorrhage Prevention
Brief Title: EMG for Uterotonic Efficiency Estimation
Acronym: EMGPHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Lucovnik, assistant professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-398/2019/7
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Postpartum Hemorrhage
Keywords: electohysterography; postpartum hemorrhage; uterine electromyography
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbetocin (Experimental): Patients will receive a single dose of carbetocin 100 mcg (Pabal ®) at admission to high dependency obstetric unit after cesarean section.
  Interventions: Drug: Carbetocin
- oxytocin (Active Comparator): Patients will receive 5 units of oxytocin ( Syntocinon ®) as a 250 ml 0.9% NaCl infusion at admission to high dependency obstetric unit after cesarean section.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Patients will receive a single dose of carbetocin 100 mcg (Pabal ®) at admission to high dependency obstetric unit after cesarean section.
  Arms: carbetocin
Drug: Oxytocin — Patients will receive 5 units of oxytocin ( Syntocinon ®) as a 250 ml 0.9% NaCl infusion at admission to high dependency obstetric unit after cesarean section.
  Arms: oxytocin

SUMMARY:
Studies found conflicting results on efficacy of uterotonic agents used to prevent and treat uterine atony, the most common cause of postpartum hemorrhage. Uterine EMG can be used to objectively assess myometrial contractility and, consequently, efficacy of different uterotonics.

The investigators are planning a single-center, randomized, open-label trial to compare uterine EMG parameters in women receiving oxytocin vs. those receiving carbetocin after cesarean delivery.

DETAILED DESCRIPTION:
RATIONALE

Postpartum hemorrhage is the leading cause of maternal mortality worldwide. In the Western world the estimated risk of life threatening postpartum hemorrhage is 2 on 1000 births. Most frequently (up to 90% of cases of postpartum hemorrhage) it is a consequence of uterine atony or inappropriate uterine contraction. In clinical practice preventing postpartum hemorrhage is key and routinely, different prophylactic uterotonic drugs are used. The first-line recommended drug for postpartum hemorrhage prevention is oxytocin. However, a recent Cochrane meta-analysis concluded that the most effective drugs (compared to oxytocin) to prevent postpartum hemorrhage of 500 ml or more are ergometrine with oxytocin, misoprostol with oxytocin and carbetocin.

Carbetocin is a synthetic heat-stable analogue of oxytocin, with a longer half-life. It shares the same mechanism of action and the same side-effects as oxytocin. The recommended dose of carbetocin is 100 μg, which is equivalent to 10 μg (5 IU) of oxytocin. In the WHO carbetocin multicenter, double-blind, randomized trial, the intramuscular administration of 100 μg of heat-stable carbetocin was discovered to be noninferior to the administration of 10 IU of oxytocin for the prevention of postpartum hemorrhage after vaginal birth. Some studies have found carbetocin to be an effective prophylactic agent with a favourable side effect profile for the third stage of labour in caesarean sections, reducing the use of additional uterotonic agents, blood and recovery time. Moreover, carbetocin was found to be effective in reducing the need for additional uterotonic use and postpartum blood transfusion in women at increased risk of postpartum hemorrhage undergoing cesarean delivery. In one study, carbetocin was also found to be more effective than oxytocin in preventing postpartum hemorrhage in twin pregnancies delivered by cesarean section.

Uterine contractions in pregnancy, labour and postpartum can be detected using electromyography. Myometrial contractility can be objectively and non-invasively assessed in vivo by monitoring uterine electromyography (EMG), as uterine contractions are the result of the electrical activity generated and propagated in the myometrium.

To our knowledge, no study has reported oxytocin or carbetocin effects using postpartum electromyography.

OBJECTIVE The objective of the study is to compare efficacy and objectively quantify the effect of carbetocin (Pabal ®) with electromyography compared to the standard uterotonic oxytocin (Syntocinon ®) for postpartum hemorrhage prevention.

METHODS Single-center, randomized, open-label trial.

After signed informed consent, the cesarean section will be performed. All the patients will receive 5 IU of oxytocin bolus and a single oxytocin infusion (10 IU). Subsequently patients will be transferred to high dependency unit and allocated randomly into one of two groups:

1. Carbetocin group Patients will receive a single dose of carbetocin 100 mcg (Pabal ®). An electromyogram of the uterus will be performed and a blood sample will be obtained. After 2-3 hours another electromyogram will follow, as well as a visual and quantified estimation of blood loss.
2. Oxytocin group Patients will receive 5 IU of oxytocin (Syntocinon ®) as a 250 ml 0.9% NaCl infusion. An electromyogram of the uterus will be performed and a blood sample will be obtained. After 2-3 hours another electromyogram will follow, as well as a visual and quantified estimation of blood loss.

Another blood sample will be routinely obtained 24 hours after the caesarean section.

Statistical analysis

From previous EMG studies, there has been reported difference in means of EMG PS peak frequency in labor vs. non-labor patients of (0.56 - 0.44 = 0.12 Hz), and a standard deviation of 0.15 Hz. Using power of 0.80, and an α - 0.05, with t-test, gives a desired sample size of 26 per group minimum.

All data will be analyzed according to a pre-established statistical plan. Statistical analyses will be performed with SPSS software (version 24.0; IBM Corporation, Armonk, New York).

Data will be entered as numerical or categorical, as appropriate. Shapiro-Wilk test will be used to assess normality of distribution. Parametric statistics will be carried out for normally distributed variables; for non-normal distribution, nonparametric statistics will be used. Data with normal distribution will be described using minimum, maximum and mean with standard deviation. Data with non-normal distribution will be shown using minimum, maximum, median, and interquartile range (IQR). Comparisons will be carried out between the study groups using independent Student's t test or Mann-Whitney U test for continuous and with Chi-square test for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with singleton pregnancies at term ( ≥37 weeks of pregnancy) scheduled for elective cesarean section after one previous cesarean section.

Exclusion Criteria:

* Contraindications for any of the study drugs.
* Anaemia Hb <100g
* History of postpartum hemorrhage
* Uterine fibroids
* Blood clotting disorder
* Placental disorder ( Placenta previa, placenta accreta)
* Preeclampsia
* Renal, cardiac or hepatic dysfunction.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Power density spectrum peak frequency of uterine EMG bursts | within 3 hours from starting treatments
  Change in Power density spectrum (PDS) peak frequency of uterine EMG bursts between EMG at admission and 2-3 hours after treatment

SECONDARY OUTCOMES:
Power density spectrum peak amplitude of uterine EMG bursts | within 3 hours from starting treatments
  Change in Power density spectrum (PDS) peak amplitude of uterine EMG bursts between EMG at admission and 2-3 hours after treatment.
Frequency and duration of uterine EMG bursts | within 3 hours from starting treatments
  Change in frequency and duration of uterine EMG bursts between EMG at admission and 2-3 hours after treatment.
Propagation velocity of uterine EMG signals | within 3 hours from starting treatments
  Propagation velocity of uterine EMG signals between EMG at admission and 2-3 hours after treatment.
Power density spectrum integral of uterine EMG bursts | within 3 hours from starting treatments
  Power density spectrum (PDS) integral of uterine EMG bursts between EMG at admission and 2-3 hours after treatment.
Change in hematocrit | within 24 hours after delivery
  Change in hematocrit between admission to high dependency unit and 24 hours after cesarean delivery.
Change in hemoglobin | within 24 hours after delivery
  Change in hemoglobin between admission to high dependency unit and 24 hours after cesarean delivery.
Quantified blood loss | within 3 hours from starting treatments
  Blood loss during treatments (from admission to the high dependency unit to EMG measurements after 2-3 hours) will be weighted.

CONTACTS AND LOCATIONS:
Overall Officials: Miha Lucovnik, MD,PhD, Study Chair — UMCL
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paljk Likar I, Becic E, Pezdirc N, Gersak K, Lucovnik M, Trojner Bregar A. Comparison of Oxytocin vs. Carbetocin Uterotonic Activity after Caesarean Delivery Assessed by Electrohysterography: A Randomised Trial. Sensors (Basel). 2022 Nov 21;22(22):8994. doi: 10.3390/s22228994. PMID 36433591